CLINICAL TRIAL: NCT03544203
Title: Multicentre Observational Study on Community Acquired Intraabdominal Infections Management: the PERICOM Study
Brief Title: Multicentre Observational Study on Community Acquired Intraabdominal Infections Management
Acronym: PERICOM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03407-46; 2017-A03407-46 (Other: ANSM)
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2019-01

CONDITIONS: Intraabdominal Infections
Keywords: intraabdominal infections; peritonitis; critically ill
MeSH Terms: conditions — Intraabdominal Infections; Peritonitis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraabdominal infection require rapid care management including antibiotic therapy and source control. Morbidity and mortality associated with Intraabdominal infections remain high. French recommendations have been edited in 2000 further updated in 2014. Delay in diagnosis and surgery can lead to worsened outcomes. However, little data are available on early community-acquired intraabdominal infections management to identify risk factors of inadequate management.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* patients admitted to emergency department for a diagnosis of proven or suspected intraabdominal infection requiring surgery

Exclusion Criteria:

* primary intraabdominal infection
* health-care associated intraabdominal infection
* abdominal trauma
* patient under guardianship
* opt out consent
* patient already enrolled in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to emergency department for a diagnosis of proven or suspected intraabdominal infection requiring surgery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
length of stay | 6 month

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU d'Amiens, Amiens, Amiens
  - AP HM La Timone, Marseille, Marseille
  - Le Kremlin-Bicêtre, Paris, Paris
  - CHU Angers, Angers
  - Hia Percy, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHU Grenoble La Tronche, Grenoble
  - CHRU Lille, Lille
  - Lyon-Sud Pierre Bénite, Lyon
  - Ap Hm La Timone, Marseille
  - CHU Nimes, Nîmes
  - CHU Bichat Claude Bernard, Paris
  - CHU Strasbourg, Strasbourg

REFERENCES:
- [Result] Roger C, Garrigue D, Bouhours G, Dupont H, Bouzat P, Bardon J, Pottecher J, Montravers P, Michelet P, Perbet S, Aymart K, Incagnoli P, Lloret S, Louart B, Harrois A; ACUTE committee. Time to source control and outcome in community-acquired intra-abdominal infections: The multicentre observational PERICOM study. Eur J Anaesthesiol. 2022 Jun 1;39(6):540-548. doi: 10.1097/EJA.0000000000001683. PMID 35608877